CLINICAL TRIAL: NCT05714371
Title: Retrospective Assessment of Adverse Events-related Healthcare Resource Utilization and Costs of Immune Checkpoint Inhibitor and Targeted Therapy for Adjuvant Treatment of Melanoma
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CTMT212AUS57
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Ipilimumab; pembrolizumab; dabrafenib; trametinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Immunotherapy (IO): Patients receiving IO
  Interventions: Drug: Nivolumab; Drug: Ipilimumab + nivolumab; Drug: Pembrolizumab
- Targeted therapy (TT): Patients receiving TT
  Interventions: Drug: Dabrafenib + trametinib

INTERVENTIONS:
Drug: Nivolumab — Patients receiving nivolumab
  Groups: Immunotherapy (IO)
Drug: Ipilimumab + nivolumab — Patients receiving ipilimumab + nivolumab
  Groups: Immunotherapy (IO)
Drug: Pembrolizumab — Patients receiving pembrolizumab
  Groups: Immunotherapy (IO)
Drug: Dabrafenib + trametinib — Dabrafenib + trametinib
  Groups: Targeted therapy (TT)

SUMMARY:
This was a retrospective cohort study using the PharMetrics database. The analysis was conducted using the most recent 5 years of data from the database, January 1, 2015, to October 30, 2020. Included patients were followed for outcome evaluation from the index date (first prescription of treatment, immunotherapy [IO], or targeted therapy [TT] following diagnosis of non-metastatic malignant melanoma and evidence of first lymph node resection), until the first occurrence or end of continuous eligibility or end of the study period.

ELIGIBILITY:
Inclusion Criteria

* Patients with at least one diagnosis of malignant melanoma of skin anytime from the start of data collection until the start of study period.
* Patients with a procedure of first lymph node dissection or nodal basin ultrasound surveillance, per the National Comprehensive Cancer Network (NCCN) guidelines version 2.2020. The first lymph node dissection / nodal basin ultrasound surveillance signified that the patient was eligible to receive systemic treatment as adjuvant therapy.
* The first lymph node dissection or nodal basin ultrasound surveillance (index adjuvant date) must have had a diagnosis of malignant melanoma of skin within 6 months, to ensure that the dissection was related to melanoma.
* Patients with at least pharmacy or medical claim for the study drugs within 1 year on and after index date. The index date was the date of first prescription of study drug, IO (i.e., nivolumab, ipilimumab + nivolumab, pembrolizumab) or dabrafenib + trametinib.
* At least 18 years of age at the time of adjuvant treatment initiation.
* Patients with at least 6 months of continuous enrollment prior to the index date.
* Patients with at least 6 months of continuous enrollment after the index date.
* If necessary, there were additional criteria of absence of secondary malignancy (including metastatic site).

Exclusion Criteria

* Patients with a diagnosis of non-melanoma primary malignancy during the 6 months pre-index period.
* Patients with chemotherapy or interferon alpha before index date.
* Patients with pregnancy any time during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study
Sampling Method: Non-Probability Sample
Enrollment: 618 (Actual)
Dates: Start 2021-10-02 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-27 (Actual)

PRIMARY OUTCOMES:
Number of patients on first systemic adjuvant therapy with adverse avents (AEs) | Up to approximately 5 years

SECONDARY OUTCOMES:
Number of patients with AEs following first systemic adjuvant therapy completion/discontinuation. | Up to approximately 5 years
Healthcare resource utilization (HCRU) associated with AEs on first systemic adjuvant therapy | Up to approximately 5 years
Healthcare costs associated with AEs on first systemic adjuvant therapy | Up to approximately 5 years
HCRU associated with AEs following first systemic adjuvant therapy completion/discontinuation | Up to approximately 5 years
Healthcare costs associated with AEs following first systemic adjuvant therapy completion/discontinuation | Up to approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States